CLINICAL TRIAL: NCT06864481
Title: Description, Course and Treatment of Immune Checkpoint Inhibitor-induced Hepatitis
Brief Title: Prospective Cohort of Immune Checkpoint Inhibitor-induced Hepatitis
Acronym: CO-CHILI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association Française pour l'Etude du Foie (AFEF) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0283
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-03

CONDITIONS: Liver Injury; Secondary to Immune Checkpoint Inhibitors; Cancer Patients
Keywords: Immune checkpoint inhibitors; Immunotherapy; Drug-induced liver injury; Hepatitis; Cholangitis; Ursodeoxycholic acid
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Hepatitis; Cholangitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immune Checkpoint Inhibitor-Induced Hepatitis: Observational cohort
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — one Blood sample (20 ml)

SUMMARY:
Background and Study Rationale Immune checkpoint inhibitors (ICI) are a breakthrough cancer treatment that boosts the immune system to fight tumors. While effective, they can cause immune-related side effects, including liver inflammation (ICI-induced hepatitis or CHILI), which affects up to 25% of patients. Severe cases requiring treatment discontinuation are rare but challenging to manage.

Study Objective This multicenter prospective study aims to better understand CHILI, its clinical patterns, treatment response, and risk of recurrence. It will focus on different types of liver injury (cholestatic, hepatocellular, or mixed) to guide better treatment decisions.

Innovation and Approach Currently, there is no clear consensus on how to manage CHILI or when to safely restart immunotherapy. This study will collect real-world data from adult patients treated with ICIs, following international guidelines or a pragmatic approach when no consensus exists. Findings will help improve care strategies for patients experiencing ICI-related liver toxicity.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years

  * Patient willing to participate in the study
  * Patient with cancer receiving neoadjuvant, adjuvant, or maintenance treatment · Patient treated with ICI, either as monotherapy or in combination with another antitumor treatment (targeted therapy, chemotherapy, or radiotherapy), either de novo or after a first-line treatment including ICIs
  * Patient who has received at least one injection of an ICI ·
  * Onset of hepatitis following treatment initiation, defined by the following criteria:

    * ALT (alanine aminotransferase) ≥ 5 times the upper normal limit
    * ALP (alkaline phosphatase) ≥ 2 times the upper normal limit
    * ALT (alanine aminotransferase) ≥ 3 times the upper normal limit and bilirubin ≥ 2 times the upper normal limit ·
  * Patient with grade 3 or 4 hepatitis, according to the current CTCAE classification
  * Exclusion criteria:
* Patient with another cause of acute hepatitis, including viral, autoimmune, ischemic, acute alcoholic hepatitis, or Wilson's disease.
* Patient unable to express their non-opposition to participate in the study.
* Person deprived of liberty, under guardianship or curatorship, or in an emergency situation.
* Person not affiliated with a social security system or without entitlement to healthcare coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be included at the hospital
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-04-22 (Estimated); Study Completion 2028-04-22 (Estimated)

PRIMARY OUTCOMES:
Ratio cholestatic phenotype, cytolytic phenotype and mixed phenotype | Day0, Day14, Day30, Day 90, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No